CLINICAL TRIAL: NCT01472926
Title: Alteplase-Tenecteplase Trial Evaluation for Stroke Thrombolysis - Pilot Phase (ATTEST)
Brief Title: Alteplase-Tenecteplase Trial Evaluation for Stroke Thrombolysis- (ATTEST)
Acronym: ATTEST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010-024541-67; TSA 2010/04 (Other Grant/Funding Number: The Stroke Association); 2010-024541-67 (EudraCT Number)
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2012-08

CONDITIONS: Stroke
Keywords: acute ischaemic stroke; stroke; thrombolysis; thrombolytic drug therapy; CT perfusion; CT angiography; brain imaging
MeSH Terms: conditions — Stroke | interventions — Tenecteplase; Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tenecteplase 0.25 mg/kg (Experimental): Intravenous tenecteplase 0.25 mg/kg (single bolus, maximum 25 mg)
  Interventions: Drug: Tenecteplase
- Alteplase 0.9 mg/kg (Active Comparator): Intravenous alteplase 0.9 mg/kg (10% bolus and 90% as IV infusion over 1 hour, maximum 90 mg)
  Interventions: Drug: alteplase

INTERVENTIONS:
Drug: Tenecteplase — Intravenous (IV) tenecteplase 0.25 mg/kg (single bolus; maximum dose 25 mg)
  Other Names: Metalyse; TNK
  Arms: Tenecteplase 0.25 mg/kg
Drug: alteplase — Intravenous alteplase 0.9mg/kg to maximum of 90mg, given as 10% bolus and 90% of dose over 1 hour infusion
  Other Names: Actilyse; recombinant tissue plasminogen activator (rtPA)
  Arms: Alteplase 0.9 mg/kg

SUMMARY:
A pilot evaluation of tenecteplase compared to alteplase in acute ischaemic stroke patients currently eligible for intravenous alteplase treatment in a prospective, randomised, blinded outcome evaluation clinical trial using brain imaging as a biomarker.

DETAILED DESCRIPTION:
Newer thrombolytic agents such as tenecteplase have pharmacological features (higher fibrin binding specificity and longer half-life) that may be advantageous when compared to older agents such as alteplase with respect to arterial recanalisation, ease of administration, and reduced bleeding risk. No other clinical trial is currently evaluating alternative thrombolytic strategies in patients who are eligible to receive standard intravenous alteplase, instead concentrating on extending the population for IV thrombolysis.

The ATTEST pilot phase will use brain imaging as a biomarker for key clinical response variables, with penumbral salvage as the primary end-point and secondary end-points including recanalisation as well as conventional clinical scales.

The findings of this study are anticipated to provide data on sample size and event rates to inform the design of a definitive, confirmatory, pragmatic, randomised, controlled trial with clinical endpoints.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of supratentorial acute ischaemic stroke with score of at least 1 on the NIH Stroke Scale
* male or non pregnant female >=18 years
* within 4.5 hours of onset as defined by time since last known well
* CT perfusion and CT Angiogram examination acquired prior to treatment

Exclusion Criteria:

* Contraindications to thrombolytic drug treatment for stroke

  * Evidence of intracranial haemorrhage or significant non-stroke intracranial pathology (including central nervous system neoplasm, aneurysm or arteriovenous malformation) on pre-treatment CT
  * Established hypodensity on pre-treatment brain CT of more than one third of the middle cerebral artery territory or Alberta Stroke Programme Early CT (ASPECT) Score <4 (sulcal effacement or loss of grey-white differentiation in cortical territories alone are not counted towards ASPECT score)
  * Hypodensity consistent with recent cerebral ischaemia other than the presenting event
  * Very severe stroke (eg NIHSS>25)
  * systolic blood pressure (BP)> 185 or diastolic BP> 110 mm Hg, or aggressive management (intravenous pharmacotherapy) necessary to reduce BP to these limits
  * If on warfarin, International Normalised Ratio (INR) <1.4
  * Current prescription of non-warfarin oral anticoagulant drugs
  * Significant abnormality of coagulation parameters pre-treatment (prolonged INR or activated partial thromboplastin time (APTT), or platelet count <100,000/mm3)
  * administration of heparin within the previous 48 hours and a thromboplastin time exceeding the upper limit of normal for laboratory, or use of therapeutic dose low molecular weight heparin within 48h
  * Clinical history suggestive of subarachnoid haemorrhage even if no blood is evident on CT
  * Risk of bleeding (Major surgery within previous 1 month; intracranial or spinal surgery; recent trauma to the head or cranium; prolonged cardiopulmonary resuscitation (> 2 minutes) within the past 2 weeks; acute pericarditis and/or subacute bacterial endocarditis; acute pancreatitis; severe hepatic dysfunction, including hepatic failure, cirrhosis, portal hypertension (oesophageal varices) and active hepatitis; active peptic ulceration; any known history of haemorrhagic stroke or stroke of unknown origin; arterial aneurysm and known arteriovenous malformation)
  * Dependent (mRS 3-5) pre-stroke
  * Blood glucose <2 mmol/l or >18 mmol/l
  * Seizure at onset of symptoms unless brain imaging identifies positive evidence of significant brain ischaemia (eg CTA confirmed arterial occlusion, early ischaemic change on plain CT, hypoperfusion on CTP)
  * Pregnancy
* Known impaired renal function (estimated Glomerular Filtration Rate <30 ml/min) precluding contrast CT
* Known allergy to radiological contrast
* History of allergies to active substances in either trial medication, or to excipients including gentamicin
* Severe concurrent medical condition that would prevent participation in study procedures (e.g. cardia failure with severe pulmonary oedema)or with life expectancy <=3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12-10 (Actual); Study Completion 2013-12-10 (Actual)

PRIMARY OUTCOMES:
Percent penumbral salvage at 24-48h (initial penumbra volume on computed tomography perfusion (CTP) imaging versus 24-48h CT infarct volume. | 48 hours
  Percent penumbral salvage at 24-48h (initial CTP-defined penumbra volume versus 24-48h CT infarct volume.

SECONDARY OUTCOMES:
Proportion of patients exhibiting recanalisation (on computed tomography angiography, CTA) 24-48 hours post treatment | 48 hours
  Proportion of patients exhibiting recanalisation (measured by CTA) 24-48 hours post treatment
Early clinical improvement 24 hours post treatment | 24 hours
  Early clinical improvement (National Institutes of Health Stroke Scale [NIHSS] score reduced by >=4 points, or = 0 or 1) 24 hours post treatment
Proportion of patients with symptomatic intracerebral haemorrhage (SICH) on 24-48 hour CT | 48 hours
  Proportion of patients with symptomatic ICH (SICH) on 24-48 hour CT:
  * by Safe Implementation of Thrombolysis Monitoring Study (SITS-MOST) definition - parenchymal haematoma type 2 (PH2/PHr2) + NIHSS deterioration by >=4 points at 24 hours
  * Any ICH
Distribution of functional outcome by modified Rankin Scale (mRS) scores at Day 30 | 30 Days
  Distribution of outcome scores on the modified Rankin Scale (mRS)
Distribution of functional outcome scores (mRS) at Day 90 | 90 days
  Distribution of functional outcome scores (mRS)
Proportion of patients with favourable clinical outcome (mRS 0-1) at Day 30 | 30 days
  Proportion of patients with favourable clinical outcome (mRS 0-1)
Proportion of patients with favourable clinical outcome (mRS 0-1) at Day 90 | 90 days
  Proportion of patients with favourable clinical outcome (mRS 0-1)
Average 'home time' by day 90 | 90 Days
  Average 'home time' (number of nights spent in non-institutional private residence) by Day 90
Mortality at Day 90 | 90 Days

CONTACTS AND LOCATIONS:
Overall Officials: Keith Muir, Study Chair — The University of Glasgow
Locations (1):
- Southern General Hospital, Glasgow, Scotland, United Kingdom

REFERENCES:
- [Derived] Bivard A, Huang X, McElduff P, Levi CR, Campbell BC, Cheripelli BK, Kalladka D, Moreton FC, Ford I, Bladin CF, Davis SM, Donnan GA, Muir KW, Parsons MW. Impact of Computed Tomography Perfusion Imaging on the Response to Tenecteplase in Ischemic Stroke: Analysis of 2 Randomized Controlled Trials. Circulation. 2017 Jan 31;135(5):440-448. doi: 10.1161/CIRCULATIONAHA.116.022582. Epub 2016 Dec 13. PMID 27965285
- [Derived] Huang X, Moreton FC, Kalladka D, Cheripelli BK, MacIsaac R, Tait RC, Muir KW. Coagulation and Fibrinolytic Activity of Tenecteplase and Alteplase in Acute Ischemic Stroke. Stroke. 2015 Dec;46(12):3543-6. doi: 10.1161/STROKEAHA.115.011290. Epub 2015 Oct 29. PMID 26514192
- [Derived] Huang X, Cheripelli BK, Lloyd SM, Kalladka D, Moreton FC, Siddiqui A, Ford I, Muir KW. Alteplase versus tenecteplase for thrombolysis after ischaemic stroke (ATTEST): a phase 2, randomised, open-label, blinded endpoint study. Lancet Neurol. 2015 Apr;14(4):368-76. doi: 10.1016/S1474-4422(15)70017-7. Epub 2015 Feb 26. PMID 25726502